CLINICAL TRIAL: NCT04017039
Title: Sleep, Blood Pressure and Vascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Christopher DeSouza, Professor, University of Colorado, Boulder
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 160646
Record Dates: First submitted 2019-07-02; First posted 2019-07-12 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Blood Pressure; Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 (No Intervention): Phase I is a cross-sectional study to compare endothelial vasodilator and fibrinolytic function in adults with elevated blood pressure who habitually sleep more than 7 hours/night (normal sleep) and those who habitually sleep less than 6.5 hr/night (short sleep)
- Phase 2 (Experimental): Phase II is an intervention study to determine the effects of individualized targeted sleep interventions that increase sleep duration and improve sleep quality on endothelial vasodilator and fibrinolytic function in adults with elevated blood pressure who habitually sleep less than 6.5 hr/night (Specific Aims 3).
  Interventions: Other: Targeted Sleep Intervention

INTERVENTIONS:
Other: Targeted Sleep Intervention
  Arms: Phase 2

SUMMARY:
The investigators hypothesize that chronic insufficient sleep is associated with diminished endothelium-dependent nitric oxide-mediated vasodilation and endothelial tissue-type plasminogen activator release in adults with elevated blood pressure. Furthermore, the investigators hypothesize that the postulated diminishment in endothelial vasodilator and fibrinolytic function with insufficient sleep will be due, at least in part, to increased oxidative stress. Furthermore, increasing sleep duration and improving sleep quality will increase both endothelium-dependent nitric oxide-mediated vasodilation and endothelial tissue-type plasminogen activator release in adults with elevated blood pressure. Increases in endothelial vasodilator and fibrinolytic function will be due, at least in part, to reduced oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be men and women of all races and ethnic backgrounds aged 45-65 years.

All women will be premenopausal, perimenopausal or post-menopausal not taking hormone replacement therapy.

Subjects will be prehypertensive/hypertensive (Stage 1 hypertension) defined as resting systolic blood pressure 125-159 mmHg and/or diastolic blood pressure 75-99 mmHg.

Subjects will have no overt signs of disease as assessed by:

1. medical history;
2. physical examination;
3. electrocardiogram and BP at rest and maximal exercise;
4. sedentary as determined from the Stanford Physical Activity Questionnaire (<35 kcal/wk) and will not have engaged in any program of regular physical activity for at least 6 months prior to the study.
5. Subjects that have a pre-existing diagnosis of obstructive sleep apnea, or are determined to have obstructive sleep apnea based on their sleep disorders screening visit will be allowed in the study, but will not take part in the sleep intervention/post sleep intervention visits.

Exclusion Criteria:

History of stroke (phone screen and medical record) Peripheral vascular disease (phone screen and medical record) History of anaphylaxis to betadine, lidocaine, iodine Body mass index > 40 kg/m2

Subjects taking blood pressure-or diabetes related medication Chronic Insomnia (prior or current diagnosis) History of or current psychiatric disorder (e.g., prior or current diagnosis, current BDI-II>13; BAI>10) Significant organ system dysfunction/disease (e.g. diabetes, severe pulmonary, kidney disease) History of seizure disorder Pregnant/nursing Positive toxicology screen-(THC, OPI, AMP, COC, PCP, BAR, BZO, MAMP/MDMA upon sleep lab admission)

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2023-05 (Actual)

PRIMARY OUTCOMES:
Phase 1: Systolic Blood Pressure (SBP) | SBP will be measured during Phase 1 at the participants week 1 visit.
Phase 2: Systolic Blood Pressure (SBP) | SBP will be measured during Phase 2 at the participants week 8 visit.
  SBP measured following the participants 8 week sleep intervention
Phase 1: Diastolic Blood Pressure (DBP) | DBP will be measured during Phase 1 at the participants week 1 visit.
Phase 2: Diastolic Blood Pressure (DBP) | DBP wwill be measured during Phase 2 at the participants week 8 visit.
  DBP measured following the participants 8 week sleep intervention
Phase 1: Forearm blood flow (FBF) response to Acetylcholine (ACh) | FBF response to ACh will be measured during Phase 1 at the participants visit 3 which is ~3 weeks from their respective start date.
Phase 2: FBF response to Acetylcholine (ACh) | FBF response to ACh will be measured during Phase 2 at the participants visit 9 which is ~13 weeks from their respective start date.
  FBF to ACh will be measured following the participants 8 week sleep intervention
Phase 1: FBF response to Sodium Nitroprusside (NTP) | FBF response to NTP will be measured during Phase 1 at the participants visit 3 which is ~3 weeks from their respective start date.
Phase 2: FBF response to Sodium Nitroprusside (NTP) | FBF response to NTP will be measured during Phase 2 at the participants visit 9 which is ~13 weeks from their respective start date.
  FBF to NTP will be measured following the participants 8 week sleep intervention
Phase 1: Endothelial t-PA Release in response to Bradykinin (BDK) | t-PA release will be measured during Phase 1 at the participants visit 3 which is ~3 weeks from their respective start date.
Phase 2: Endothelial t-PA Release in response to Bradykinin (BDK) | t-PA release will be measured during Phase 2 at the participants visit 9 which is ~13 weeks from their respective start date.
  Endothelial t-PA release will be measured following the participants 8 week sleep intervention.
Phase 1: FBF response to L-NMMA | FBF response to L-NMMA will be measured during Phase 1 at the participants visit 3 which is ~3 weeks from their respective start date.
Phase 2: FBF response to L-NMMA | FBF response to L-NMMA will be measured during Phase 2 at the participants visit 9 which is ~13 weeks from their respective start date.
  FBF to L-NMMA will be measured following the participants 8 week sleep intervention.
Phase 1: FBF response to ACh+L-NMMA | FBF response to ACh+L-NMMA will be measured during Phase 1 at the participants visit 3 which is ~3 weeks from their respective start date.
Phase 2: FBF response to ACh+L-NMMA | FBF response to ACh+L-NMMA will be measured during Phase 2 at the participants visit 9 which is ~13 weeks from their respective start date.
  FBF to ACh+L-NMMA will be measured following the participants 8 week sleep intervention

SECONDARY OUTCOMES:
Phase 1: Pittsburgh Sleep Quality Index (PSQI) | The PSQI questionnaire will be administered during Phase 1 at the participants week 1 visit.
  This questionnaire assesses sleep quality. Scores range from 0 indicating no difficulty and 21 indicating severe difficulty.
Phase 2: PSQI | The PSQI questionnaire will be administered during Phase 2 at the participants week 8 visit.
  This questionnaire assesses sleep quality. Scores range from 0 indicating no difficulty and 21 indicating severe difficulty.
Phase 1: Insomnia Severity Index | The insomnia severity index questionnaire will be administered during Phase 1 at the participants week 1 visit.
  This questionnaire is used to assess the nature and severity of insomnia. Scores range from 0 no insomnia to 28 severe insomnia.
Phase 2: Insomnia Severity Index | The insomnia severity index questionnaire will be administered during Phase 2 at the participants week 8 visit.
  This questionnaire is used to assess the nature and severity of insomnia. Scores range from 0 no insomnia to 28 severe insomnia.
Phase 1: Epworth Sleepiness Scale | The Epworth Sleepiness scale questionnaire will be administered during Phase 1 at the participants week 1 visit.
  This questionnaire is used to assess daytime sleepiness. Scores range from 0 normal daytime sleepiness to 24 severe daytime sleepiness.
Phase 2: Epworth Sleepiness Scale | The Epworth Sleepiness scale questionnaire will be administered during Phase 2 at the participants week 8 visit.
  This questionnaire is used to assess daytime sleepiness. Scores range from 0 normal daytime sleepiness to 24 severe daytime sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher DeSouza, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- UC-Boulder Clinical and Translational Research Center, Boulder, Colorado, United States